CLINICAL TRIAL: NCT00300274
Title: A 24-month, Multi-center, Randomized, Open-label, Non-inferiority Study of Efficacy and Safety Comparing Two Exposures of Concentration-controlled Everolimus With Reduced Cyclosporine Versus 3.0 g Mycophenolate Mofetil With Standard Dose Cyclosporine in de Novo Heart Transplant Recipients
Brief Title: Efficacy and Safety of Everolimus in Recipients of Heart Transplants to Prevent Acute and Chronic Rejection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2310
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-07

CONDITIONS: Graft Rejection
Keywords: Everolimus; heart transplant; heart disease; transplantation; heart IVUS assessment at 12 months; rate of graft loss; acute rejection episodes; survival
MeSH Terms: conditions — Heart Diseases | interventions — Everolimus; Mycophenolic Acid; Cyclosporine; Adrenal Cortex Hormones

ARMS (3):
- everolimus 1.5 mg (Experimental): Within 72 hours after transplantation participants received 0.75 mg everolimus tablets twice a day 12 hours apart for a total 1.5 mg daily dose in combination with reduced cyclosporine and standard dose corticosteroids for 24 months. The everolimus dose could be adjusted to maintain a target everolimus trough level of 3-8 ng/mL.
  Interventions: Drug: everolimus; Drug: cyclosporine; Drug: corticosteroids
- everolimus 3.0 mg (Experimental): Within 72 hours after transplantation participants received 1.5 mg everolimus tablets twice a day 12 hours apart for a total 3.0 mg daily dose in combination with reduced cyclosporine and standard dose corticosteroids for 24 months. The everolimus dose could be adjusted to maintain a target everolimus trough level of 6-12 ng/mL.
  Randomization of new patients in this arm was prematurely stopped as of 27 March 2008 due to high mortality rate, as per Data Monitoring Committee.
  Interventions: Drug: everolimus; Drug: cyclosporine; Drug: corticosteroids
- mycophenolate mofetil (Active Comparator): Within 72 hours after transplantation participants received 3 tablets 500 mg mycophenolate mofetil twice a day 12 hours apart for a total daily dose of 3000 mg in combination with a standard cyclosporine dose and standard dose corticosteroids for 24 months.
  Interventions: Drug: mycophenolate mofetil; Drug: cyclosporine; Drug: corticosteroids

INTERVENTIONS:
Drug: everolimus — Everolimus supplied as 0.75 mg tablets. Everolimus was also supplied in 0.25 mg and 0.5 mg tablets for dose adjustments.
  Other Names: Zortress®; Certican®
  Arms: everolimus 1.5 mg; everolimus 3.0 mg
Drug: mycophenolate mofetil — Mycophenolate mofetil supplied as 500 mg tablets.
  Other Names: Cellcept®
  Arms: mycophenolate mofetil
Drug: cyclosporine — Cyclosporine reduced dose in the everolimus arms (approximately half of the standard dose) and standard dose in the mycophenolate mofetil arm.
  Other Names: Neoral®
Drug: corticosteroids — Corticosteroids standard dose.

SUMMARY:
This trial was to examine the impact of everolimus and reduced dose of cyclosporine on efficacy and safety compared to mycophenolate mofetil and a standard dose of cyclosporine in heart transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cardiac recipients 18-70 years of age undergoing primary heart transplantation.
* The graft must be functional at time of randomization.

Exclusion Criteria:

* Patients who are recipients of multiple solid organ transplants or tissue transplants or have previously received organ transplants.
* Patients who are recipients of ABO incompatible transplants.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2006-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (64):
- United States (26):
  - UCLA Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford U Sch, Falk Cardiovasular Research Ctr., Stanford, California
  - University of Florida Shands Hospital, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Loyola Univerisity Medical School, Maywood, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Recanati Miller Transplant Institute, New York, New York
  - UNC Division of Cardiology, Chapel Hill, North Carolina
  - Duke University Heart Failure Research, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiovascular Consultants, Austin, Texas
  - University of Texas Medical Branch, Div of Cardio Thoracic, Galveston, Texas
  - Methodist Hospital/DeBakey Heart Failure Research Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Wisconsin - Madison Medical School, Madison, Wisconsin
  - St. Luke's Medical Center Cardiac Services, Milwakee, Wisconsin
- Argentina (2):
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Fundacion Favalaro, Buenos Aires
- Australia (3):
  - St Vincents Hospital, Darlinghurst, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Perth Hospital, Perth, Western Australia
- Universitaet Wien, Vienna, Austria
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - St Paul's Hospital, Vancouver, British Columbia
  - New Halifax Infirmary, Halifax, Nova Scotia
  - Toronto General Hospital, Toronto, Ontario
  - Institut Univ. de cardiologie et pneumologie de Quebec, Sainte-Foy, Quebec
- France (5):
  - Hopital Cardiologique de Lyon, Lyon
  - Hopital Georges Pompidou, Paris
  - Hopital Pitie Salpetriere, Paris
  - CHU de Strasbourg Hopital Civil Medicale B, Strasbourg
  - CHU Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Herz- u. Diabeteszentrum NRW/Ruhr-Univ. Bochum, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Kliniken der Med. Hochschule, Hanover
  - Universitaetsklinikum Kiel, Kiel
  - Universitaetsklinik Regensburg, Regensburg
- Italy (6):
  - Az. Osp. di Bologna Policl. S. Orsola-Malpighi Univ. degli Studi, Bologna
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - A.O.-Universita di Padova-Universita degli Studi, Padua
  - Fodazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Ospedaliera S. Camillo-Forlanini, Roma
  - Az. Ospedaliero-Universitaria S. Giovanni Battista di Torino, Torino
- Auckland Hospital, Auckland, New Zealand
- Rikshospitalet, Hjertemedisinskavdeling, Oslo, Norway
- Cardiovascular Center of Puerto Rico and the Caribbean, San Juan, Puerto Rico
- Spain (2):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Puerta de Hierro Majadahonda, Madrid
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Papworth Hospital, Cambridge
  - Wythenshawe Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus 1.5 mg: Within 72 hours after transplantation participants received 0.75 mg everolimus tablets twice a day 12 hours apart for a total 1.5 mg daily dose in combination with reduced cyclosporine and standard corticosteroids for 24 months. The everolimus dose could be adjusted to maintain a target everolimus trough level of 3-8 ng/mL.
- Everolimus 3.0 mg: Within 72 hours after transplantation participants received 1.5 mg everolimus tablets twice a day 12 hours apart for a total 3.0 mg daily dose in combination with reduced cyclosporine and standard dose corticosteroids for 24 months. The everolimus dose could be adjusted to maintain a target everolimus trough level of 6-12 ng/mL.
Period: Overall Study
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Started | 282 | 168 | 271
Completed 12 Month | 250 | 149 | 248
Completed | 236 | 141 | 226
Not Completed | 46 | 27 | 45
Not completed — Withdrawal by Subject | 12 | 3 | 14
Not completed — Lost to Follow-up | 3 | 4 | 5
Not completed — Death | 31 | 20 | 25
Not completed — Re-transplant | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil | Total
Number analyzed (Participants) | 282 | 168 | 271 | 721
Age Continuous [Mean (Standard Deviation); unit: years] | 51.1 (10.99) | 48.9 (12.06) | 50.2 (11.88) | 50.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 39 | 51 | 147
  Male | 225 | 129 | 220 | 574

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Efficacy Failure at 12 Months
Description: Composite efficacy failure was defined as Biopsy Proven Acute Rejection(BPAR) of International Society for Heart and Lung Transplantation(ISHLT) grade ≥3A, Acute Rejection associated with Hemodynamic Compromise, Graft loss/Retransplant, Death or Loss to follow-up.
  Identification of acute rejection was based on the local pathologist's evaluation of endomyocardial biopsy slides.
  Hemodynamic compromise was present if 1 or more of the following were met: Ejection fraction ≤30% or 25% lower than Baseline or Fractional shortening ≤20% or 25% lower than Baseline and/or use of inotropic treatment.
Time Frame: 12 Months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 282 | 168 | 271
Percentage of participants | 35.1 | 35.1 | 33.6

2. Secondary Outcome: Percentage of Participants With Graft Loss/Re-transplant, Death or Loss to Follow-up at 12 Months
Description: Loss to follow-up for this composite endpoint included participants who did not experience graft loss/re-transplant or death and whose last day of contact was prior to Day 316 (start day of the Month 12 visit window).
Time Frame: 12 Months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 282 | 168 | 271
Percentage of participants | 11.7 | 11.9 | 8.9

3. Secondary Outcome: Renal Function Measured by Glomerular Filtration Rate (GFR) at 12 Months
Description: GFR was calculated using the Modification of Diet and Renal Disease (MDRD) formula:
  GFR [mL/min/1.73m^2] = 186.3*(C^-1.154)*(A^-0.203)*G*R where C is the serum concentration of creatinine [mg/dL] A is age [years] G=0.742 when gender is female, otherwise G=1 R=1.21 when race is black, otherwise R=1
Time Frame: 12 Months
Population: Participants from the intent-to-treat population (all randomized participants) with data available for analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73^2
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 241 | 141 | 238
mL/min/1.73^2 | 59.21 (23.113) | 59.78 (23.141) | 64.37 (28.365)

4. Secondary Outcome: Change From Baseline in the Average Maximum Intimal Thickness at Month 12
Description: Maximum intimal thickness was assessed using Intravascular Ultrasound (IVUS). IVUS is a technique for taking ultrasound pictures of the wall of an artery from inside the artery itself. It shows the thickness of the artery wall and any narrowing of the artery.
Time Frame: Baseline, Month 12
Population: IVUS population consisted of randomized patients who had a minimum of 11 matched slices between IVUS images from Baseline and from Month 12 (IVUS Centers).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 88 | 37 | 101
mm | 0.03 (0.052) | 0.04 (0.06) | 0.07 (0.110)

5. Secondary Outcome: Percentage of Participants With Cardiac Allograft Vasculopathy (CAV) at Month 12
Description: Cardiac allograft vasculopathy is defined as a 0.5 mm increase in maximum intimal thickness as measured by Intravascular Ultrasound (IVUS) in at least one matched slice between baseline and Month 12.
Time Frame: 12 Months
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 88 | 37 | 101
Percentage of participants | 12.5 | 21.6 | 26.7

6. Secondary Outcome: Percentage of Participants With Biopsy-proven Acute Rejection (BPAR of ISHLT Grade ≥ 3A), Acute Rejection Associated With Hemodynamic Compromise (HDC), Graft Loss/Re-transplant and Death at Month 12
Description: Identification of acute rejections was based on the local pathologist's evaluation of endomyocardial biopsy slides.
  Hemodynamic compromise was present if 1 or more of the following were met: Ejection fraction ≤ 30% or 25% lower than Baseline or Fractional shortening ≤ 20% or 25% lower than Baseline, and/or use of inotropic treatment.
Time Frame: 12 Months
Population: Intent-to-treat population includes all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 282 | 168 | 271
Percentage of participants
  AR associated with HDC | 3.9 | 3.0 | 2.6
  BPAR of ISHLT ≥ 3A | 22.3 | 25.6 | 24.7
  Death | 7.8 | 10.1 | 4.8
  Graft loss/re-transplant | 1.4 | 3.0 | 1.8

7. Secondary Outcome: Percentage of Participants With Composite Efficacy Failure at 24 Months
Description: Composite efficacy failure was defined as Biopsy Proven Acute Rejection (BPAR) of International Society for Heart and Lung Transplantation grade ≥ 3A, Acute Rejection associated with Hemodynamic Compromise, Graft loss/Retransplant, Death or Loss to follow-up.
  Identification of acute rejections was based on the local pathologist's evaluation of endomyocardial biopsy slides.
  Hemodynamic compromise was present if 1 or more of the following were met: Ejection fraction ≤ 30% or 25% lower than Baseline or Fractional shortening ≤ 20% or 25% lower than Baseline and/or use of inotropic treatment.
Time Frame: 24 Months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 282 | 168 | 271
Percentage of participants | 39.4 | 41.1 | 41.3

8. Secondary Outcome: Percentage of Participants With Graft Loss/Re-transplant, Death or Loss to Follow-up at 24 Months
Description: Loss to follow-up for this composite endpoint included participants who did not experience graft loss/re-transplant or death and whose last day of contact was prior to Day 631 (start day of 24 Month visit window).
Time Frame: 24 Months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 282 | 168 | 271
Percentage of participants | 15.2 | 16.1 | 15.1

9. Secondary Outcome: Renal Function Calculated by Glomerular Filtration Rate (GFR) at 24 Months
Description: GFR was calculated using the Modification of Diet and Renal Disease (MDRD) formula:
  GFR [mL/min/1.73m^2] = 186.3*(C^-1.154)*(A^-0.203)*G*R
  C is the serum concentration of creatinine [mg/dL] A is age [years] G=0.742 when gender is female, otherwise G=1 R=1.21 when race is black, otherwise R=1
Time Frame: 24 Months
Population: Participants from the intent-to-treat population (all randomized participants) with data available for analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73^2
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 227 | 132 | 127
mL/min/1.73^2 | 59.50 (22.438) | 61.84 (25.247) | 64.52 (23.764)

10. Secondary Outcome: Percentage of Participants With Biopsy-proven Acute Rejection (BPAR of ISHLT Grade ≥ 3A), Acute Rejection (AR) Associated With Hemodynamic Compromise (HDC), Graft Loss/Re-transplant and Death at Month 24
Description: Identification of acute rejections was based on the local pathologist's evaluation of endomyocardial biopsy slides.
  Hemodynamic compromise was present if 1 or more of the following were met: Ejection fraction ≤ 30% or 25% lower than Baseline or Fractional shortening ≤ 20% or 25% lower than Baseline, and/ or use of inotropic treatment.
Time Frame: 24 Months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Number analyzed (Participants) | 282 | 168 | 271
Percentage of participants
  AR associated with HDC | 4.3 | 3.6 | 5.2
  BPAR of ISHLT grade ≥ 3A | 24.1 | 28.6 | 27.3
  Death | 10.6 | 11.9 | 9.2
  Graft loss/re-transplant | 2.5 | 3.0 | 3.7

ADVERSE EVENTS:
Arm/Group | Everolimus 1.5 mg | Everolimus 3.0 mg | Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 209/279 | 119/167 | 168/268
Other Adverse Events (participants affected / at risk) | 275/279 | 165/167 | 262/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 1.5 mg (N=279) | Everolimus 3.0 mg (N=167) | Mycophenolate Mofetil (N=268)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 4 | 2 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 7 | 3 | 10
Atrial flutter (Cardiac disorders) | 4 | 1 | 5
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 2
Atrial thrombosis (Cardiac disorders) | 0 | 2 | 2
Atrioventricular block (Cardiac disorders) | 0 | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 5 | 3
Cardiac failure (Cardiac disorders) | 1 | 1 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 4 | 1 | 4
Cardiac perforation (Cardiac disorders) | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 5 | 3 | 4
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 1 | 6
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Dilatation atrial (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 0 | 2
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0
Nodal rhythm (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 5 | 0 | 4
Pericardial cyst (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 38 | 18 | 12
Pericardial haemorrhage (Cardiac disorders) | 1 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 2 | 0
Pericarditis constrictive (Cardiac disorders) | 2 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 2 | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 2 | 3 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 1
Sinus arrest (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 3
Tricuspid valve incompetence (Cardiac disorders) | 3 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 2
Ventricular asystole (Cardiac disorders) | 1 | 0 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 1
Retinal artery thrombosis (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 2 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 4 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 0
Ileitis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4 | 7
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 3 | 5
Asthenia (General disorders) | 3 | 0 | 1
Cardiac death (General disorders) | 0 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 3 | 4 | 2
Concomitant disease progression (General disorders) | 1 | 0 | 0
Crepitations (General disorders) | 1 | 0 | 0
Device breakage (General disorders) | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 6
Feeling hot (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 2 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 2 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 2
Malaise (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 6 | 3 | 5
Non-cardiac chest pain (General disorders) | 8 | 2 | 3
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 6 | 5 | 4
Pyrexia (General disorders) | 12 | 14 | 10
Sudden cardiac death (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 2 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Allergy to animal (Immune system disorders) | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 1
Heart transplant rejection (Immune system disorders) | 20 | 13 | 26
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Transplant rejection (Immune system disorders) | 2 | 1 | 2
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 1
Abscess neck (Infections and infestations) | 0 | 0 | 1
Acute pulmonary histoplasmosis (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1 | 0
Aspergillosis (Infections and infestations) | 2 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 2 | 1
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 2 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 2
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 1 | 2
Candida pneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 2
Cerebral aspergillosis (Infections and infestations) | 0 | 0 | 2
Chlamydial infection (Infections and infestations) | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 2 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 2
Cytomegalovirus gastritis (Infections and infestations) | 0 | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 3 | 5 | 10
Cytomegalovirus syndrome (Infections and infestations) | 0 | 0 | 3
Cytomegalovirus viraemia (Infections and infestations) | 1 | 2 | 8
Device related infection (Infections and infestations) | 2 | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 0 | 1
Enterobacter pneumonia (Infections and infestations) | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1 | 0
Fungal abscess central nervous system (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Fungal peritonitis (Infections and infestations) | 1 | 0 | 0
Fungal sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 1 | 4
Gastroenteritis viral (Infections and infestations) | 3 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 3
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1 | 0
Infected lymphocele (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1
Intraspinal abscess (Infections and infestations) | 0 | 1 | 0
Listeriosis (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 5 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 1 | 0
Mediastinitis (Infections and infestations) | 4 | 1 | 2
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1 | 0
Mycobacterium chelonei infection (Infections and infestations) | 0 | 0 | 1
Myocarditis mycotic (Infections and infestations) | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 3 | 2
Pericarditis fungal (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 2 | 0
Pneumonia (Infections and infestations) | 15 | 11 | 8
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 3
Pneumonia escherichia (Infections and infestations) | 2 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 1 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 3 | 1 | 1
Pneumonia primary atypical (Infections and infestations) | 2 | 1 | 2
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Post procedural pneumonia (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 5 | 5 | 2
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1
Pseudomonas bronchitis (Infections and infestations) | 0 | 0 | 1
Purulent pericarditis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyothorax (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1
Salmonella sepsis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 7 | 6 | 2
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Septic embolus (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 4 | 3 | 2
Sinusitis (Infections and infestations) | 3 | 2 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0
Spinal cord infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal mediastinitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 3 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 1
Urinary tract infection (Infections and infestations) | 5 | 0 | 5
Urosepsis (Infections and infestations) | 1 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 3 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 5 | 0 | 1
Wound infection (Infections and infestations) | 1 | 2 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Complications of transplanted heart (Injury, poisoning and procedural complications) | 2 | 0 | 2
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of sternum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 2 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 | 0 | 4
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 4 | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 1
Atrial pressure increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 2 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Catheterisation cardiac (Investigations) | 0 | 1 | 0
Cells in urine (Investigations) | 0 | 0 | 1
Central venous pressure increased (Investigations) | 1 | 0 | 0
Culture wound positive (Investigations) | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 2 | 2
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 0 | 0
Immunosuppressant drug level (Investigations) | 1 | 0 | 0
Immunosuppressant drug level decreased (Investigations) | 0 | 0 | 1
Immunosuppressant drug level increased (Investigations) | 1 | 1 | 0
Left ventricular end-diastolic pressure increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1
Sputum culture positive (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 6 | 6 | 6
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 4
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 2 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 2
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 2 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 4 | 1 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 2 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Hemiparesis (Nervous system disorders) | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 2
Migraine (Nervous system disorders) | 1 | 2 | 1
Neurological symptom (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 2
Polyneuropathy (Nervous system disorders) | 2 | 1 | 4
Sciatica (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 5 | 1 | 6
Thalamic infarction (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 3 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 2
Delirium (Psychiatric disorders) | 0 | 2 | 1
Depression (Psychiatric disorders) | 1 | 1 | 2
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 3
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 | 0
Nephrosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 10 | 0 | 3
Renal failure acute (Renal and urinary disorders) | 12 | 13 | 13
Renal failure chronic (Renal and urinary disorders) | 1 | 2 | 0
Renal impairment (Renal and urinary disorders) | 3 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Colpocele (Reproductive system and breast disorders) | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 4 | 6
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Incisional drainage (Surgical and medical procedures) | 0 | 1 | 0
Angiodysplasia (Vascular disorders) | 1 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2 | 3
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 2 | 0 | 1
Haemodynamic instability (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 4 | 2 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 5 | 4
Intermittent claudication (Vascular disorders) | 1 | 0 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 1 | 0
Lymphocele (Vascular disorders) | 5 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 0
Lymphorrhoea (Vascular disorders) | 1 | 0 | 0
Malignant hypertension (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 2
Phlebitis (Vascular disorders) | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 1.5 mg (N=279) | Everolimus 3.0 mg (N=167) | Mycophenolate Mofetil (N=268)
Anaemia (Blood and lymphatic system disorders) | 105 | 60 | 74
Leukocytosis (Blood and lymphatic system disorders) | 37 | 27 | 27
Leukopenia (Blood and lymphatic system disorders) | 36 | 29 | 67
Neutropenia (Blood and lymphatic system disorders) | 8 | 4 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 25 | 25
Atrial fibrillation (Cardiac disorders) | 20 | 13 | 22
Left ventricular hypertrophy (Cardiac disorders) | 16 | 5 | 12
Mitral valve incompetence (Cardiac disorders) | 15 | 7 | 18
Palpitations (Cardiac disorders) | 12 | 14 | 14
Pericardial effusion (Cardiac disorders) | 93 | 51 | 69
Sinus tachycardia (Cardiac disorders) | 13 | 9 | 7
Tachycardia (Cardiac disorders) | 20 | 14 | 23
Tricuspid valve incompetence (Cardiac disorders) | 28 | 17 | 24
Abdominal distension (Gastrointestinal disorders) | 11 | 8 | 17
Abdominal pain (Gastrointestinal disorders) | 29 | 17 | 26
Abdominal pain upper (Gastrointestinal disorders) | 17 | 9 | 17
Constipation (Gastrointestinal disorders) | 70 | 42 | 63
Diarrhoea (Gastrointestinal disorders) | 62 | 43 | 67
Dyspepsia (Gastrointestinal disorders) | 17 | 9 | 16
Nausea (Gastrointestinal disorders) | 64 | 52 | 72
Vomiting (Gastrointestinal disorders) | 33 | 21 | 45
Asthenia (General disorders) | 16 | 12 | 21
Chills (General disorders) | 12 | 12 | 13
Fatigue (General disorders) | 39 | 22 | 50
Non-cardiac chest pain (General disorders) | 38 | 10 | 26
Oedema peripheral (General disorders) | 133 | 69 | 119
Pyrexia (General disorders) | 47 | 22 | 38
Heart transplant rejection (Immune system disorders) | 6 | 2 | 15
Bronchitis (Infections and infestations) | 7 | 7 | 15
Cytomegalovirus infection (Infections and infestations) | 14 | 7 | 25
Herpes zoster (Infections and infestations) | 8 | 4 | 23
Nasopharyngitis (Infections and infestations) | 35 | 12 | 32
Oral candidiasis (Infections and infestations) | 10 | 3 | 14
Oral herpes (Infections and infestations) | 7 | 9 | 15
Upper respiratory tract infection (Infections and infestations) | 34 | 16 | 32
Urinary tract infection (Infections and infestations) | 18 | 19 | 20
Incision site pain (Injury, poisoning and procedural complications) | 20 | 19 | 20
Post procedural discharge (Injury, poisoning and procedural complications) | 14 | 6 | 7
Procedural pain (Injury, poisoning and procedural complications) | 35 | 24 | 32
Blood creatinine increased (Investigations) | 25 | 17 | 18
Blood triglycerides increased (Investigations) | 13 | 9 | 7
Cytomegalovirus test positive (Investigations) | 4 | 9 | 18
Haemoglobin decreased (Investigations) | 19 | 6 | 22
Weight increased (Investigations) | 14 | 5 | 15
White blood cell count decreased (Investigations) | 11 | 12 | 35
Decreased appetite (Metabolism and nutrition disorders) | 10 | 11 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 20 | 8 | 22
Fluid overload (Metabolism and nutrition disorders) | 47 | 30 | 43
Gout (Metabolism and nutrition disorders) | 15 | 6 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 38 | 22 | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 32 | 21 | 31
Hyperkalaemia (Metabolism and nutrition disorders) | 34 | 17 | 34
Hyperlipidaemia (Metabolism and nutrition disorders) | 22 | 9 | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 41 | 23 | 30
Hypoglycaemia (Metabolism and nutrition disorders) | 15 | 10 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 39 | 25 | 32
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 | 20 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 13 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 51 | 17 | 42
Muscle spasms (Musculoskeletal and connective tissue disorders) | 41 | 21 | 36
Muscular weakness (Musculoskeletal and connective tissue disorders) | 19 | 6 | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 | 4 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 9 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 11 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 9 | 25
Dizziness (Nervous system disorders) | 37 | 19 | 27
Headache (Nervous system disorders) | 85 | 39 | 70
Paraesthesia (Nervous system disorders) | 23 | 10 | 17
Tremor (Nervous system disorders) | 58 | 33 | 60
Anxiety (Psychiatric disorders) | 41 | 22 | 35
Depression (Psychiatric disorders) | 27 | 14 | 26
Insomnia (Psychiatric disorders) | 77 | 32 | 60
Renal failure (Renal and urinary disorders) | 44 | 25 | 27
Renal impairment (Renal and urinary disorders) | 23 | 8 | 13
Erectile dysfunction (Reproductive system and breast disorders) | 16 | 6 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 15 | 7 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 67 | 23 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 25 | 47
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 13 | 9 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 9 | 16
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 65 | 37 | 57
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 15 | 4 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 | 5 | 10
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 18
Acne (Skin and subcutaneous tissue disorders) | 23 | 18 | 28
Hirsutism (Skin and subcutaneous tissue disorders) | 8 | 9 | 6
Rash (Skin and subcutaneous tissue disorders) | 15 | 17 | 17
Hypertension (Vascular disorders) | 132 | 72 | 125
Hypotension (Vascular disorders) | 23 | 13 | 27
Jugular vein thrombosis (Vascular disorders) | 14 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.